CLINICAL TRIAL: NCT00337441
Title: Chronic Anemia And Fatigue In Elderly Patients: A Randomized Double-Blind Placebo-Controlled Cross-Over Study With Epoetin Alfa.
Brief Title: Treatment of Chronic Anemia With Epoetin Alfa in Elderly
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Research and Education Foundation of Michael Reese Hospital (Other)
Collaborators: Ortho Biotech Clinical Affairs, L.L.C. (Industry); Cook County Health (Other Government); Mercy Hospital and Medical Center, Illinois (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PR02-32-031
Record Dates: First submitted 2006-06-14; First posted 2006-06-16 (Estimated); Last update posted 2006-06-16 (Estimated); Status verified 2006-06

CONDITIONS: Anemia
Keywords: Chronic Anemia; Anemia; Chronic Diseases; Elderly; Epoetin alfa; Fatigue; Quality of life; Mobility
MeSH Terms: conditions — Anemia; Chronic Disease; Fatigue | interventions — Epoetin Alfa; Pharmaceutical Preparations

INTERVENTIONS:
Drug: Epoetin Alfa (drug)

SUMMARY:
The purpose of this study is to determine if chronic anemia can be corrected with epoetin alfa and does the subsequent correction lead to an improvement in fatigue,quality of life or mobility among elderly.

DETAILED DESCRIPTION:
Chronic Anemia is common among elderly. Given their somewhat non-specific nature, the clinical symptoms of anemia are often difficult to attribute directly to the anemia itself. However, it is known that anemic older adults are at an increased risk of mortality, disability, higher risk of falls, poorer quality of life, worsening cognitive function, increase hospitalization risk, and increased healthcare utilization than their non-anemic counterparts.

Yet so far, there have been no treatment studies to demonstrate the benefits of correction of chronic anemia.

Epoetin Alfa (Procrit) is a manufactured form of a naturally occurring hormone that is given as an injection by a medical professional to stimulate the bone marrow's production of red blood cells.

This study is to explore, can chronic anemia be corrected with epoetin alfa and does the subsequent correction lead to an improvement in fatigue, quality of life or mobility among elderly.

Overall this is a 32 week treatment study.

In this study, participants with chronic anemia will receive either Epoetin alfa or placebo (saline injection) under the skin for 16 weeks. After 16 weeks the participants who were receiving epoetin will be switched to placebo and those who were receiving placebo earlier will go on now to receive epoetin alfa for 16 weeks.

At the end of 32 weeks we will compare, if epoetin alfa corrected the anemia, how individuals felt in respect to their fatigue levels, quality of life and did mobility improve during the study.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older Diagnosed with chronic anemia Hemoglobin level less than or equal to 11.5 g/dl Community dwelling Able to make monthly clinic visits

Exclusion Criteria:

* Currently on Epoetin alfa or similar preparations Having nutritional anemia Having active cancer or received recent treatment for cancer On treatment for Kidney disease Diagnosis of dementia Inability to ambulate

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 62
Dates: Start 2003-01; Study Completion 2005-07

PRIMARY OUTCOMES:
Hemoglobin
Fatigue
Quality of Life

SECONDARY OUTCOMES:
Quality of Life
Mobility

CONTACTS AND LOCATIONS:
Overall Officials: Parag Agnihotri, Principal Investigator — Research and Education Foundation of Michael Reese
Locations (2):
- United States (2):
  - John H. Stroger Jr. Hospital of Cook County, Chicago, Illinois
  - Mercy Hospital and Medical Center, Chicago, Illinois

REFERENCES:
- [Background] Guralnik JM, Eisenstaedt RS, Ferrucci L, Klein HG, Woodman RC. Prevalence of anemia in persons 65 years and older in the United States: evidence for a high rate of unexplained anemia. Blood. 2004 Oct 15;104(8):2263-8. doi: 10.1182/blood-2004-05-1812. Epub 2004 Jul 6. PMID 15238427
- [Background] Weiss G, Goodnough LT. Anemia of chronic disease. N Engl J Med. 2005 Mar 10;352(10):1011-23. doi: 10.1056/NEJMra041809. No abstract available. PMID 15758012
- [Background] Penninx BW, Pahor M, Cesari M, Corsi AM, Woodman RC, Bandinelli S, Guralnik JM, Ferrucci L. Anemia is associated with disability and decreased physical performance and muscle strength in the elderly. J Am Geriatr Soc. 2004 May;52(5):719-24. doi: 10.1111/j.1532-5415.2004.52208.x. PMID 15086651
- [Background] Cella D, Zagari MJ, Vandoros C, Gagnon DD, Hurtz HJ, Nortier JW. Epoetin alfa treatment results in clinically significant improvements in quality of life in anemic cancer patients when referenced to the general population. J Clin Oncol. 2003 Jan 15;21(2):366-73. doi: 10.1200/JCO.2003.02.136. PMID 12525531